CLINICAL TRIAL: NCT02179606
Title: A Multi-Center, Randomized, Subject and Evaluator Blind, Split-Face Comparative Medical Device Clinical Study to Evaluate the Efficacy and Safety of Dermalax Implant Plus to Restylane® Sub-Q for Correction of Nasolabial Folds
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Dermalax Implant Plus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Across Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC-13-01
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-03

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Dermalax Implant Plus (Experimental): Subject injected in the nasolabial folds of one side of the face in the initial treatment period.
  Interventions: Device: Dermalax Implant Plus; Device: Restylane Sub-Q
- Restylane Sub-Q (Active Comparator): Subject injected in the nasolabial folds of one side of the face in the initial treatment period.
  Interventions: Device: Dermalax Implant Plus; Device: Restylane Sub-Q

INTERVENTIONS:
Device: Dermalax Implant Plus — Dermalax implant plus injection into one nasolabial fold(NFL) of one side of the face(blinded, split-face study design) in the initial treatment period.
Device: Restylane Sub-Q — Restylane Sub-Q injection into one nasolabial fold(NFL) of one side of the face(blinded, split-face study design) in the initial treatment period.

SUMMARY:
This study is to verify that Dermalax Implant Plus is not inferior to the reference device, Restylane® Sub-Q, in terms of efficacy and safety in the correction of nasolabial folds

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects no younger than 30 and no more than 75 years of age.
2. Subjects who scored 3 or 4 on the Wrinkle Severity Rating Scale (WSRS) and want to improve the appearance of their nasolabial folds (the subject does not need to have the same score on both sides.*)

   *The scores need not to be same on both sides, but the two nasolabial folds should have symmetry in the range of 3-4.
3. Subjects who have symmetric nasolabial folds.

Exclusion Criteria:

1. Subjects who received an antithrombotic agent within 2 weeks prior to screening (with the exception of low dose Aspirin less than 300 mg/day)
2. Subjects who have a history of bleeding disorder.
3. Subjects who have received calcium hydroxyapatite, CaHA injection in nasolabial area.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement of wrinkle severity system scale(WSRS) scores of both Dermalax implant plus and Restylane® Sub-Q Group | baseline, week 12
  Improvement of wrinkle severity system scale(WSRS) scores at week 12 compared to baseline by independent evaluator using photos.

SECONDARY OUTCOMES:
Improvement of wrinkle severity system scale(WSRS) scores of both Dermalax implant plus and Restylane® Sub-Q Group | baseline, at week 2~24
  Improvement of wrinkle severity system scale(WSRS) scores at week2, week8, week 16, week 24 compared to baseline by independent evaluator using photos.
Proportion of subjects whose Global Aesthetic improvement Scale (GAIS) scores improved | at week 2~24
  Proportion of subjects whose Global Aesthetic improvement Scale (GAIS) scores improved at week2, week 8, week 12, week 16, week 24 evaluated by investigator at site
100 mm visual analogue scale (VAS) scores evaluation | week 0
  100 mm visual analogue scale (VAS) scores at both nasolabial folds evaluated by subjects at application of the devices

OTHER OUTCOMES:
Safty evaluation | for 24weeks
  adverse events, laboratory test, physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Beom Joon Kim, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Jong Hoon Lee, MD, Principal Investigator — Eulji General Hospital
Locations (2):
- South Korea (2):
  - Chung-ang University Hospital, Seoul
  - Eulji General Hospital, Seoul